CLINICAL TRIAL: NCT05782816
Title: Low-Dose Versus High-Dose Oxytocin Dosing for Induction and Augmentation of Labor: A Randomized Control Trial
Brief Title: Low-Dose Versus High-Dose Oxytocin Dosing for Induction and Augmentation of Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-0240
Record Dates: First submitted 2023-02-21; First posted 2023-03-24 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Labor Long
Keywords: induction of labor; augmentation of labor; oxytocin; pitocin; high dose; mode of delivery
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose oxytocin (Active Comparator): The low dose oxytocin group will receive a controlled infusion pump at a proximal port on the peripheral IV line. The infusion will start at 2 milli-units/min and will be increased by 2 milli-units/min every 20 minutes. Maximum rate of infusion is 40 milli-units/min. Oxytocin infusion rate is adjusted to maintain adequate uterine contractions.
  Interventions: Drug: Oxytocin (Low dose)
- High dose oxytocin (Active Comparator): The high dose oxytocin group will receive a controlled infusion pump at a proximal port on the peripheral IV line. The infusion will start at 6 milli-units/min and will be increased by 6 milli-units/min every 20 minutes. Maximum rate of infusion is 40 milli-units/min. Oxytocin infusion rate is adjusted to maintain adequate uterine contractions.
  Interventions: Drug: Oxytocin (High dose)

INTERVENTIONS:
Drug: Oxytocin (Low dose) — Low dose oxytocin
  Other Names: Pitocin; Syntocinon
  Arms: Low dose oxytocin
Drug: Oxytocin (High dose) — High dose oxytocin
  Other Names: Pitocin; Syntocinon
  Arms: High dose oxytocin

SUMMARY:
The goal of this clinical trial is to compare oxytocin infusion rates for induction and augmentation of labor in nulliparous women. The main question[s] it aims to answer are:

* Does a high dose oxytocin infusion protocol affect length of induction to delivery interval?
* Does a high dose oxytocin infusion protocol affect mode of delivery?
* Does a high dose oxytocin infusion protocol affect maternal and neonatal outcomes?

Participants will be randomized to either low- or high-dose oxytocin groups:

* The low dose group will receive an infusion to start at 2 milli-units/min and will be increased by 2 milli-units/min every 20 minutes. The maximum rate of infusion is 40 milli-units/min.
* The high dose group will receive an infusion to start at 6 milli-units/min and will be increased by 6 milli-units/min every 20 minutes. Maximum rate of infusion is 40 milli-units/min.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 years old
* Singleton gestation
* Nulliparous
* Vertex presentation
* Gestational age greater than or equal to 37 weeks
* No prior uterine surgery
* Presents for elective or medically indicated induction of labor
* Need for augmentation of labor with oxytocin

Exclusion Criteria:

* Previous cervical ripening using non-mechanical methods
* Patient unable or unwilling to provide verbal consent
* Contraindications to vaginal delivery
* Fetal demise or life-limiting anomaly
* Allergy to oxytocin
* Non-reassuring fetal heart tracing prior to inclusion
* Maternal pulmonary edema prior to inclusion
* Fetal growth restriction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 170 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wang, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Oxytocin: The low dose oxytocin group will receive a controlled infusion pump at a proximal port on the peripheral IV line. The infusion will start at 2 milli-units/min and will be increased by 2 milli-units/min every 20 minutes. Maximum rate of infusion is 40 milli-units/min. Oxytocin infusion rate is adjusted to maintain adequate uterine contractions.
  Oxytocin: Low dose oxytocin
- High Dose Oxytocin: The high dose oxytocin group will receive a controlled infusion pump at a proximal port on the peripheral IV line. The infusion will start at 6 milli-units/min and will be increased by 6 milli-units/min every 20 minutes. Maximum rate of infusion is 40 milli-units/min. Oxytocin infusion rate is adjusted to maintain adequate uterine contractions.
  Oxytocin: High dose oxytocin
Period: Overall Study
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Started | 85 | 85
Completed | 84 | 85
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin | Total
Number analyzed (Participants) | 84 | 85 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 85 | 169
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Age measured in years.
  years | 24.0 [18 to 40] | 23.8 [18 to 38] | 23.9 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants by sex at baseline.
  Participants
    Female | 84 | 85 | 169
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Number of participants by ethnicity (Hispanic or Latino / Not Hispanic or Latino) as defined by NIH/OMB standards.
  Participants
    Hispanic or Latino | 62 | 59 | 121
    Not Hispanic or Latino | 22 | 26 | 48
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery
Description: Induction to delivery time interval
Time Frame: Through delivery, on average 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
minutes | 1041.8 (537.5) | 971.1 (519.0)

2. Secondary Outcome: Mode of Delivery
Description: Vaginal or cesarean delivery
Time Frame: Through delivery, on average 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants
  vaginal delivery | 58 | 52
  cesarean delivery | 25 | 1
  operative vaginal delivery | 1 | 32

3. Secondary Outcome: Rate of Primary Cesarean Delivery
Description: Number of participants with primary cesarean delivery.
Time Frame: Through delivery, on average 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 25 | 1

4. Secondary Outcome: Maximum Dose of Oxytocin Infusion
Description: The highest oxytocin infusion rate administered to a participant during the study period.
Time Frame: Through delivery, on average 24 hours
Measure: Number; unit: mU/min
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
mU/min | 11.8 | 15.6

5. Secondary Outcome: Rate of Uterine Tachysystole
Description: The number of participants with and without fetal heart rate changes and the need for cessation or decrease in oxytocin dosage.
Time Frame: Through delivery, on average 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 15 | 22

6. Secondary Outcome: Number of Participants With Postpartum Hemorrhage
Time Frame: From delivery through the postpartum period (average duration approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 1 | 4

7. Secondary Outcome: Rate of Placental Abruption
Description: The number of participants with placental abruption.
Time Frame: Through delivery, on average 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Nausea/Vomiting Requiring Antiemetics and Diarrhea
Time Frame: From delivery (average duration approximately 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 0 | 0

9. Secondary Outcome: Rate of Maternal Infection (Endometritis, Chorioamnionitis)
Description: The number of participants with maternal maternal infections (endometritis, choriomnionitis)
Time Frame: Through delivery, on average 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 29 | 30

10. Secondary Outcome: Rate of Serious Maternal Morbidity and Mortality
Description: The number of participants with uterine rupture, admission to ICU, and septicemia or mortality.
Time Frame: Through delivery, on average 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 0 | 0

11. Secondary Outcome: Number of Neonates With One or More of: Perinatal Death, Severe Respiratory Distress Requiring Ventilation, Neonatal Encephalopathy, Neonatal Seizure, Neonatal Sepsis, 5-minute APGAR Score <7, Umbilical Artery Acidemia, Neonatal ICU Admission
Time Frame: From birth through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 7 | 10

12. Secondary Outcome: Number of Participants With Neonatal Sepsis (Confirmed With Cultures)
Time Frame: From birth through 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 0 | 0

13. Secondary Outcome: Rate of Umbilical Artery Acidemia (Base Excess <12)
Description: Number of participants with umbilical artery acidemia (base excess <12).
Time Frame: Through delivery, on average 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
Number analyzed (Participants) | 84 | 85
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Through delivery, on average 24 hours
Arm/Group | Low Dose Oxytocin | High Dose Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/85
Other Adverse Events (participants affected / at risk) | 0/84 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT05782816/Prot_SAP_000.pdf